CLINICAL TRIAL: NCT01406613
Title: A 2-year Observational Study of Bone Density and Bone Turnover After Prior Treatment With Alendronate, Ibandronate and Risedronate for Postmenopausal Osteoporosis in Secondary Care
Brief Title: Resolution of Effect of Bisphosphonates on Bone in Postmenopausal Osteoporosis
Status: Completed | Type: Observational
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: University of Sheffield (Other)
Responsible Party: Sponsor
Other Study IDs: STH15387
Record Dates: First submitted 2011-07-29; First posted 2011-08-01 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Postmenopausal Osteoporosis
Keywords: Observational; Bone Density; alendronate; ibandronate; risedronate; postmenopausal; osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A venous blood sample will be collected from each participant at each visit to analyse biochemical bone markers, and basic biochemistry analysis for eligibility screening.
  Two urine samples will be collected from each participant at each study visit, one collected on the morning prior to the study visit and a second sample on the morning of the study visit.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Particpants of previous TRIO study: All participants to this study are being observed as a follow up to a previous study which involved 4 arms. All participants to this follow up study will be subject to identical study procedures.
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — In this study we will examine the changes in bone density by DXA and QUS and bone turnover after stopping Bisphosphonate treatment. As we wish to measure the speed of offset of effects of treatment we have scheduled visits at 24 week intervals in order to fully assess this effect.

SUMMARY:
This is a 2year observational study that will recruit patients who have previously completed a randomised, open label, parallel, single centre study (TRIO Study) of three bisphosphonates: alendronate, ibandronate and risedronate. These drugs are the most commonly used group of treatments for postmenopausal osteoporosis in the UK. However, the length of time for which these treatments continue to work after they are stopped has not been fully elucidated. Without this information it is unclear as to how long doctors should treat and whether it would be good practice to give drug 'holidays'.

The investigators plan to compare the effects on bone quantity and quality of stopping these licensed bisphosphonates in patients who have taken the medication for a duration of two years. The investigators aim to recruit up to 100 postmenopausal and up to 100 premenopausal (reference range) subjects. Measurements collected at the final visit of the previous study will be used for 'baseline' values for this study.

The postmenopausal group will have an initial study visit to secure informed consent, and then further study visits at 24, 48, 72 and 96 weeks after stopping medication. Visit procedures will include:

Blood and urine samples for measurements of bone biomarkers Bone Mineral Density of the spine, hip, whole body, forearm Dual-emission X-ray absorptiometry (DXA), and heel dual X-ray and Laser (DXL) Quantitative Ultrasound of Bone (QUS) Vertebral Fracture Assessment (VFA).

The premenopausal group will have one study visit, 96 weeks after completing the previous study. Visit procedures will include:

Blood and urine samples for measurements of bone biomarkers Bone Mineral Density of the spine and hip (DXA)

A subgroup of 50 premenopausal women will also have the following measurements:

Bone Mineral Density of the whole body, forearm (DXA), and heel (DXL) Quantitative Ultrasound of Bone (QUS).

DETAILED DESCRIPTION:
The current study is an observational study aiming to compare the effects of stopping medication on bone quantity and quality, in patients who have previously taken bisphosphonate drugs for a duration of two years.

This study will recruit participants who have previously completed the TRIO study. The TRIO study aimed to compare the effects of three licensed bisphosphonates on bone quantity and quality. Participants in the treatment group of the TRIO study were randomised to treatment with one of three licensed bisphosphonates (alendronate, ibandronate and risedronate) for a duration of two years.

Measurements taken at the final TRIO study visit will be used as 'baseline' values for this study. The postmenopausal group will have an informed consent visit, followed by further study visits at 24, 48, 72 and 96 weeks after stopping medication.

Study visit procedures for the postmenopausal group will include:

Blood and urine samples for measurements of bone biomarkers at 24, 48, 72 and 96 weeks off treatment.

This study will recruit participants who have previously completed the TRIO study. The TRIO study aimed to compare the effects of three licensed bisphosphonates on bone quantity and quality. Participants in the treatment group of the TRIO study were randomised to treatment with one of three licensed bisphosphonates (alendronate, ibandronate and risedronate) for a duration of two years.

Measurements taken at the final TRIO study visit will be used as 'baseline' values for this study. The postmenopausal group will have an informed consent visit, followed by further study visits at 24, 48, 72 and 96 weeks after stopping medication.

Study visit procedures for the postmenopausal group will include:

Blood and urine samples for measurements of bone biomarkers at 24, 48, 72 and 96 weeks off treatment Height and weight at 48 and 96 weeks off treatment. Bone Mineral Density of the whole body, spine, hip, forearm (DXA) and heel (DXL) at 48 and 96 weeks off treatment Vertebral Fracture Assessment (VFA) at 48 and 96 weeks off treatment. Quantitative Ultrasound of Bone (QUS) of the heel at 48 and 96 weeks off treatment.

Participants will be given a diary at their first study visit, to record any newly prescribed medications, hospitalisations, etc. The diary will be reviewed at each study visit to record any adverse events or concomitant medications. Participants will also be asked to complete the standard Metabolic Bone Centre questionnaire at their first and final study visit, so that any changes in lifestyle can be captured. We will maintain the patients on treatment with calcium and vitamin D supplements throughout the study as this would be consistent with standard clinical practice.

The TRIO study recruited a group of premenopausal women in order to collect data to act as a reference range for the physical measurements and also to act as internal controls for the study. This study plans to recruit these control participants to continue to act as a reference range in this study.

The premenopausal group will have a single study visit, scheduled 96 weeks after completing the TRIO study. Study visit procedures for the premenopausal (reference) group will include:

Blood and urine samples for measurements of bone biomarkers Urine based pregnancy test Height and weight Bone Mineral Density of the hip and spine (DXA).

A subgroup of 50 premenopausal (reference) women will also have the following:

Bone Mineral Density of the whole body, forearm (DXA) and heel (DXL) Quantitative Ultrasound of Bone (QUS) of the heel Participants will be asked to complete the standard Metabolic Bone Centre questionnaire, so that any changes in lifestyle can be captured. Participants will also be asked about any hospitalisations, newly prescribed medications, etc to capture any adverse events and concomitant medications.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for postmenopausal women

* female be at least 7 years postmenopausal but less than 87 years of age
* be ambulatory
* be able and willing to participate in the study and provide written informed consent.
* have taken a bisphosphonate for 2 years as a participant in the TRIO study and be compliant > 80%
* have a Bone Mineral Density (BMD) T score > -2.5 at the femoral neck

Inclusion Criteria for premenopausal women

* be able and willing to participate in the study and provide written informed consent
* have previously taken part as premenopausal controls in the TRIO study
* be in good general health as determined by past medical and physical history
* be bisphosphonate naive; premenopausal women.

Exclusion Criteria:

Exclusion Criteria for postmenopausal women:

* An incident vertebral fracture or more than 5%/year bone loss at the spine or hip during the 2-year TRIO study
* Evidence of a clinically significant organic disease which could prevent the patient from completing the study, including diabetes
* Abuse of alcohol or use of illicit drugs or who consumed more than 4 units of any alcoholic beverage one day prior to the visit (i.e. subjects who might be binge drinkers)
* A history of cancer within the past 5 years excluding skin cancer non melanomas
* A history of ongoing conditions or diseases known to cause abnormalities of calcium metabolism or skeletal health (secondary osteoporosis)
* Chronic renal disease (as defined by a creatinine clearance of ≤ 30ml/min)
* Acute or chronic hepatic disease
* Malabsorption syndromes
* Hyperthyroidism as manifested by Thyrotrophin-stimulating hormone (TSH) outside the lower limit of the normal range
* Hyperparathyroidism
* Hypocalcemia or hypercalcemia
* Osteomalacia
* Cushing's syndrome
* Current use of glucocorticoid therapy
* A serum calcium less than 2.2 mmol/l and a Parathyroid hormone (PTH) above 75ng/l
* A history of any known condition that would interfere with the assessment of Dual-emission X-ray absorptiometry (DXA) at either lumbar spine or femoral neck
* Markedly abnormal clinical laboratory parameters that are assessed as clinically significant by the principal investigator
* Require, in the opinion of the consulting physician, continuation of bisphosphonate therapy.

Exclusion Criteria for premenopausal women:

* Are pregnant or nursing (lactating)
* Use of any hormonal forms of contraception/ therapy within the past 2 years that would, in the opinion of the consulting physician, affect bone metabolism.
* Use of anabolic agents such as steroids or PTH, or any bisphosphonate within the past 2 years.
* Have any history of cancer within the past 5 years. Relatively benign skin malignancies, such as basal cell carcinoma or squamous cell carcinoma, are not an exclusion if the patient has been in remission for at least 6 months prior to enrolment.
* Have any chronic disease (HIV or AIDs, clinically significant renal or cardiovascular disease, hyperthyroidism, diabetes, hyperlipidemia) or menstrual cycle irregularity (by history)).
* Have any metabolic bone disease, such as osteoporosis, Paget 's disease, osteogenesis imperfecta, or serious illness affecting normal bone homeostasis (by history and physical exam if required)
* Significant use of any medications known to affect bone metabolism (such as Phenytoin or other anticonvulsants, Selective Estrogen Receptor Modulators (SERMs), heparin or systemic glucocorticosteroids) within the past 2 years.
* Have suffered a fracture within the last 12 months
* Have anorexia nervosa, suspected bulimia (by history or physical) or obvious malnutrition
* Have a history of alcoholism, or who have consumed more than 4 units of any alcoholic beverage one day prior to the visit (i.e., subjects who might be binge drinkers)
* Have previously participated in active therapy clinical trials within the last 3 months

Max Age: 87 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants of previous TRIO study - women who either received treatment with alendronate, ibandronate and risedronate for postmenopausal osteoporosis in secondary care. Control premenopausal women will also be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2010-03 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Eastell, Professor, Principal Investigator — University of Sheffield
Locations (1):
- Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, South Yorks, United Kingdom